CLINICAL TRIAL: NCT07238946
Title: Prevalence of Musculoskeletal Pain and Its Association With Perceived Stress Among Medical Students of Pakistan: a Cross-sectional Study
Brief Title: Musculoskeletal Pain and Its Association With Stress in Medical Students
Status: Completed | Type: Observational
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Arfa Umer, Dr, Services Institute of Medical Sciences, Pakistan
Other Study IDs: MSKPainStressMed2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Muskuloskeletan Pain; Stress (Psychology)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical students: Medical students enrolled in medical colleges of Pakistan participating in a cross sectional survey assesing musculoskeletal pain and associated factors
  Interventions: Other: Observational assessment only

INTERVENTIONS:
Other: Observational assessment only — This study is purely observational. Participants will complete a questionnaire regarding musculoskeletal pain. No interventions, treatments, or procedures are administered as part of the study.

SUMMARY:
The goal of this observational study is to learn about the prevalence of musculoskeletal pain in undergraduate medical students and its association with perceived stress. The main question it aims to answer is:

Is there any association between musculoskeletal pain and stress in medical students of Pakistan? Participants filled out an online survey questions about their pain frequency and stress experienced.

DETAILED DESCRIPTION:
the study is a cross sectional study conducted in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate medical students enrolled in MBBS in medical colleges of Pakistan.

Students present during the data collection period.

Exclusion Criteria:

* Students with a previously diagnosed musculoskeletal disorder (e.g., arthritis, lupus, fibromyalgia) Incomplete questionnaire responses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of medical students enrolled at private and public medical colleges of PAKISTAN, including both males and females from all academic years. Students currently enrolled and providing informed consent are eligible. Students with pre-existing musculoskeletal disorders or those unwilling to participate are excluded
Sampling Method: Non-Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of musculoskeletal pain among medical students, assessed using a standardized questionnaire (Nordic Musculoskeletal Questionnaire). | Single assessment during academic year 2025
  Musculoskeletal pain was assessed using a validated questionnaire to determine prevalence and anatomical distribution among participants

SECONDARY OUTCOMES:
Association between stress levels and musculoskeletal pain | Single assessment during academic year 2025
  Stress level was measured using a validated scale ( Perceived Stress Scale) and analyzed for correlation with the presence, severity, and distribution of musculoskeletal pain among participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of participants, IPD will not be shared with other organizations